CLINICAL TRIAL: NCT00399841
Title: Spinal Cord Stimulation (SCS) for Neuropathic Pain of Back or Lower Extremity: A Comparison of Electrode Placement at T7 and T8
Brief Title: Spinal Cord Stimulation (SCS) for Neuropathic Pain of Back or Lower Extremity
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Investigator Resigned
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: SCS0306
Record Dates: First submitted 2006-11-13; First posted 2006-11-15 (Estimated); Results first posted 2020-12-19 (Actual); Last update posted 2020-12-19 (Actual); Status verified 2020-11

CONDITIONS: Intractable Neuropathic Pain; Pain; Back Pain; Lower Extremity Pain
Keywords: Pain; Chronic Pain; Neurostimulation
MeSH Terms: conditions — Pain; Back Pain; Chronic Pain | interventions — Spinal Cord Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Stimulation will occur at the T7 followed by T8 during the trial implant period
  Interventions: Device: Precision for Spinal Cord Stimulation
- 2 (Active Comparator): Stimulation will occur at the T8 followed by T7 during the trial implant period
  Interventions: Device: Precision for Spinal Cord Stimulation

INTERVENTIONS:
Device: Precision for Spinal Cord Stimulation — During Trial Implant Period, stimulation from single lead initially turned on at the T7 or T8 level, then crossover. At time of permanent implant, subject chooses which level they want the stimulator turned on.

SUMMARY:
The primary objective of this study is to compare the efficacy and patient preference for spinal cord stimulation (SCS) using the Precision device with the electrode array placed at T7 versus placement at T8. Eligible patients will have chronic intractable pain in the back or lower extremities and will have independently elected SCS as the next line of therapy. There is some anecdotal evidence that the coverage of the paresthesia resulting from T7 placement is preferable to that obtained by the more commonly used T8 placement but there has been no study to support this observation.

DETAILED DESCRIPTION:
The conventional implantation of the spinal cord stimulator calls for dual percutaneous leads placed at T8-T9 vertebral levels. Recently published studies as outlined in a letter to the editor of Neuromodulation suggest that a "well placed single lead will generally perform better than a dual lead." Furthermore, anecdotal reports suggest that lead placement at T7 will capture axial back pain with greater success compared to lead placement at alternative sites.

This study aims to achieve better pain treatment and paresthesia coverage by placing a single lead at T7.

ELIGIBILITY:
Inclusion Criteria:

* Be diagnosed with chronic intractable neuropathic pain of moderate to severe intensity of the back or lower extremity and meeting the criteria for post-laminectomy syndrome, be eligible for SCS, and have independently elected SCS as next line of therapy.
* Be 18 years of age or older.
* Be willing and able to comply with all study related procedures and visits.
* Be capable of reading and understanding patient information materials and giving written informed consent.

Exclusion Criteria:

* Have sensory loss in the low back or lower extremity as the primary complaint.
* Have any significant medical condition that is likely to interfere with study procedures or likely to confound evaluation of study endpoints.
* Have participated in any investigational drug or device trial in the last 4 weeks or plan to participate in any other study during the year.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2006-11 (Actual); Primary Completion 2008-05 (Actual); Study Completion 2008-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roshini Jain, Study Director — Boston Scientific Neuromodulation Corporation
Locations (1):
- Anesthesia Associates of Belleville, Belleville, Illinois, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Study: Stimulation at T7 followed by T8 or stimulation at T8 followed by T7 during the trial implant period
  Precision for Spinal Cord Stimulation: During Trial Implant Period, stimulation from single lead initially turned on at the T7 or T8 level, then crossover. At time of permanent implant, subject chooses which level they want the stimulator turned on.
- Stimulation at T7 Followed by T8: Stimulation at T7 followed by T8 during the trial implant period
  Precision for Spinal Cord Stimulation: During Trial Implant Period, stimulation from single lead initially turned on at the T7 or T8 level, then crossover. At time of permanent implant, subject chooses which level they want the stimulator turned on.
- Stimulation at T8 Followed by T7: Stimulation at T8 followed by T7 during the trial implant period
  Precision for Spinal Cord Stimulation: During Trial Implant Period, stimulation from single lead initially turned on at the T7 or T8 level, then crossover. At time of permanent implant, subject chooses which level they want the stimulator turned on.
Period: Overall Study
Arm/Group | Study | Stimulation at T7 Followed by T8 | Stimulation at T8 Followed by T7
Started | 13 | 0 (# of participants unknown. Efforts were made to locate data. No data are available) | 0 (# of participants unknown. Efforts were made to locate data. No data are available)
Permanent Implant | 6 | 0 (# of participants unknown. Efforts were made to locate data. No data are available) | 0 (# of participants unknown. Efforts were made to locate data. No data are available)
12-week | 2 | 0 (# of participants unknown. Efforts were made to locate data. No data are available) | 0 (# of participants unknown. Efforts were made to locate data. No data are available)
Completed | 1 | 0 (# of participants unknown. Efforts were made to locate data. No data are available) | 0 (# of participants unknown. Efforts were made to locate data. No data are available)
Not Completed | 12 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Insufficient data collected
Groups:
- Baseline: Enrolled subjects
Arm/Group | Baseline
Number analyzed (Participants) | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 5
  >=65 years | 8
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 3
Region of Enrollment [Number; unit: participants]
  United States | 13

OUTCOME MEASURES:

1. Primary Outcome: The Primary Efficacy Endpoint is Pain Severity After Trial Stimulation.
Time Frame: End of trial (approximately 5 days)
Population: The study was terminated and efforts were made to locate data. No study data are available
Groups:
- Stimulation at T7: Stimulation will occur at the T7 during the trial implant period
  Precision for Spinal Cord Stimulation: During Trial Implant Period, stimulation from single lead initially turned on at the T7 or T8 level, then crossover. At time of permanent implant, subject chooses which level they want the stimulator turned on.
- Stimulation at T8: Stimulation will occur at the T8 level during the trial implant period
  Precision for Spinal Cord Stimulation: During Trial Implant Period, stimulation from single lead initially turned on at the T7 or T8 level, then crossover. At time of permanent implant, subject chooses which level they want the stimulator turned on.
Arm/Group | Stimulation at T7 | Stimulation at T8
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected from enrollment through end of study (52 weeks post-activation or withdrawal).
Description: Insufficient data collected. The study was terminated and efforts were made to locate data. Number of participants/randomization assignment unknown.
Groups:
- Study: Stimulation will occur at T7 followed by T8 or T8 followed by T7 during the trial implant period
  Precision for Spinal Cord Stimulation: During Trial Implant Period, stimulation from single lead initially turned on at the T7 or T8 level, then crossover. At time of permanent implant, subject chooses which level they want the stimulator turned on.
Arm/Group | Study
All-Cause Mortality (participants affected / at risk) | 1/13
Serious Adverse Events (participants affected / at risk) | 2/13
Other Adverse Events (participants affected / at risk) | 0/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Study (N=13)
(General disorders) | 1 (2)
Twitching (Nervous system disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Insufficient data collected to report results

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes